CLINICAL TRIAL: NCT01831167
Title: Effect of Dynamic Light Application on Performance of ICU Nurses
Acronym: Tefflon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeroen Bosch Ziekenhuis (Other)
Responsible Party: Principal Investigator, K.S. Simons, MD, Jeroen Bosch Ziekenhuis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IC-JBZ-Tefflon
Record Dates: First submitted 2013-04-04; First posted 2013-04-15 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Sustained Selective Attention; Divided Attention
Keywords: dynamic light application; sustained attention; divided attention; nursing
MeSH Terms: interventions — Dynamic Light Scattering

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- dynamic light (Experimental): dynamic light
  Interventions: Other: dynamic light
- reference (No Intervention): normal light

INTERVENTIONS:
Other: dynamic light
  Arms: dynamic light

SUMMARY:
In two sessions of four days nurses will be exposed to dynamic lighting and normal (reference) lighting. Through the psychological tests T.O.D.A. (Test or divided attention) and T.O.S.S.A. (Test of sustained selective attention), then the focus tested. These two tests run both 5 times. The investigators also ask to fill out: 3 questionnaires, fatigue and mood, sleep and Questions of Life.

ELIGIBILITY:
ICU nurses working 32 hours/week or more

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
score on Test of Divided Attention | march 2013
  divided attention
Test on Sustained Selective Attention(TOSSA) | to april 2013

CONTACTS AND LOCATIONS:
Overall Officials: Koen Simons, MD, Principal Investigator — Jeroen Bosch Ziekenhuis
Locations (1):
- Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, Netherlands